CLINICAL TRIAL: NCT07066956
Title: Impacto Del Exoesqueleto Infantil Atlas 2030 en la Funcionalidad de la Marcha y en la Calidad de Vida de Niños Con Parálisis Cerebral Infantil o Patologías Afines
Brief Title: Impact of the Atlas 2030 Pediatric Exoskeleton on Gait Functionality and Quality of Life in Children With Cerebral Palsy or Related Conditions
Status: Completed | Type: Observational
Sponsor: FIDMAG Germanes Hospitalàries (Other)
Collaborators: Hospital Aita Menni (Unknown); ASPACE Gipuzkoa (Unknown)
Responsible Party: Principal Investigator, JOSE IGNACIO QUEMADA UBIS, Director Médico, FIDMAG Germanes Hospitalàries
Other Study IDs: PS2023001
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy Infantile
Keywords: Cerebral Palsy; Gait; Pediatric; Exoskeleton
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 2-14 years with cerebral palsy: Children aged 2-14 years with cerebral palsy with Gross Motor Function Classification System (GMFCS) level III, IV or V.
  They underwent intensive training with 4 weekly sessions during 6 weeks with the ATLAS 2030 exoskeleton, a wearable device that provides gait assistance through eight degrees of freedom, four for each leg, including hip, knee, and ankle rotations. During training sessions, participants were fitted with the exoskeleton and performed 25 minutes of automatic forward walking, 15 minutes of active forward walking, 15 minutes of automatic forward walking, 5 minutes of automatic backward walking, 5 minutes of active backward walking, and exoskeleton removal. During the walk, therapeutic activities based on therapeutic objectives were carried out according to the participants' abilities.
  Interventions: Device: ATLAS 2030 Exoskeleton

INTERVENTIONS:
Device: ATLAS 2030 Exoskeleton — They underwent intensive training with 4 weekly sessions during 6 weeks with the ATLAS 2030 exoskeleton, a wearable device that provides gait assistance through eight degrees of freedom, four for each leg, including hip, knee, and ankle rotations. During training sessions, participants were fitted with the exoskeleton and performed 25 minutes of automatic forward walking, 15 minutes of active forward walking, 15 minutes of automatic forward walking, 5 minutes of automatic backward walking, 5 minutes of active backward walking, and exoskeleton removal. During the walk, therapeutic activities based on therapeutic objectives were carried out according to the participants' abilities.

SUMMARY:
Title of the Study IMPACT OF THE ATLAS 2030 PEDIATRIC EXOSKELETON ON GAIT FUNCTIONALITY AND QUALITY OF LIFE IN CHILDREN WITH CEREBRAL PALSY OR RELATED CONDITIONS

Justification Cerebral palsy and gait rehabilitation It is estimated that around 93 million children worldwide have some form of moderate or severe disability. Cerebral palsy (CP) is the most common motor disability in children, with a prevalence of 1.8 per 1,000 live births in Europe. CP causes severe motor dysfunction, sometimes resulting in the inability to stand or walk. This is due to damage in areas of the central nervous system (CNS) that control movement and posture. CP causes a series of signs and symptoms such as spasticity, muscle contractures, incoordination, loss of selective motor control, or weakness, which interfere with motor function and daily living activities in these children.

As part of physical therapy, there are different types of pediatric robotic devices that assist with gait. These include: Lokomat, a stationary treadmill-based device; the G-EO System, which is also stationary and has a stair-climbing function; Innowalk, which enables standing; and other similar devices like NX-A3, Robogait, and Walkbot-K. Also notable is Prodrobot, which differs from the above as it performs suspended walking.

Walking has been shown to have physiological and functional benefits, including the prevention of muscle contractures, maintenance of bone density, and improvement of cardiovascular function. Booth et al., in their meta-analysis, suggest that gait therapy produces more beneficial effects in children with CP than conventional therapy. Moreover, effective and functional mobility-whether independent or aided by support systems-enhances children's abilities to interact with and explore their surroundings. In the treatment of neuromuscular diseases (NMDs), low-impact exercise and supported ambulation are highly beneficial.

Robot-assisted gait rehabilitation involves integrating these electromechanical systems into treatment programs. Calderón et al. argue that robotic devices enable early gait retraining and that their benefits lie in increasing training volume while reducing fatigue for both the patient and therapists. This allows for more repetitions, consistency, and quality of treatments in a safe manner.

Medical Device Description The ATLAS 2030 exoskeleton is a robotic active orthosis with 8 degrees of freedom, classified as a THKAFO-type device. It aims to improve the user's motor level, with the goal of not only increasing life expectancy but also reducing or delaying complications associated with disease progression or prolonged sitting.

It is attached to the human body in a non-invasive manner without direct skin contact, using a physical interface based primarily on straps and braces. Its chassis is adjustable in length and width for children between 100 cm and 130 cm in height.

It performs human walking with active mobility in a three-dimensional space, providing controlled movement in the sagittal and frontal planes. In addition to walking forward and backward, it replicates sit-to-stand and stand-to-sit movements.

The ATLAS exoskeleton is optimized for children with neuromuscular diseases (spinal muscular atrophy, muscular dystrophies, myopathies, etc.) and cerebral palsy. The device also self-adjusts to the patient's strength and mobility needs thanks to ARES technology, which absorbs joint disturbances and ensures safe control of the exoskeleton.

ATLAS 2030 evolves intelligently with rehabilitation progress. It is easily adjustable to the child's growth and can be put on in just 5 minutes.

Main Objective

To evaluate improvements in motor functions related to gait with the use of the ATLAS 2030 pediatric exoskeleton. Specifically, the following will be assessed:

* Gross motor function
* Range of motion in the lower limbs
* Strength in various muscle groups of the neck, trunk, and limbs
* Spasticity in the limbs
* Increase in gait capacity

Study Design Observational study under routine clinical practice with pre-, post-, and follow-up measurements

Target Disease or Disorder Inability or severe difficulty with independent walking in children aged 2 to 14 years with disabilities due to cerebral palsy or related conditions

Primary Outcome Measures

* Gross Motor Function Measure (GMFM-66): Assesses gross motor function, defined as the number of motor activities the child can perform
* 6-Minute Walk Test (6MWT): Measures the maximum distance the child can walk in six minutes, evaluated while using the exoskeleton

Study Population and Total Number of Patients 20 children between the ages of 2 and 14, with Gross Motor Function Classification System levels III, IV, or V

Treatment Duration 6 weeks of treatment and an additional 6 weeks of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy diagnosis
* Gross Motor Function Classification System (GMFCS) III, IV or V.

Exclusion Criteria:

* None

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy aged 2-14 years.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure scale (GMFMS-88) | 12 weeks
  The scale contains 88 items on a 4-point scale (0-3) that are divided into five dimensions: A) Lying and Rolling (17 items); B) Sitting (20 items); C) Crawling and Kneeling (14 items); D) Standing (13 items); and E) Walking, Running, and Jumping (24 items). A higher score on the scale indicates better gross motor function and, therefore, greater achievement of motor development milestones.

SECONDARY OUTCOMES:
6-minute walk test | 12 weeks
  It measures the distance walked in 6 minutes, with the aim of evaluating physical endurance during exercise. In this case, it was performed while using the device in active mode, forward, and threshold 1.
Total steps in active mode forward and backward | 12 weeks
  Total steps in active mode forward and backward, to measure adaptation to exercise, in this case, walking with the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospitalarioak Fundazioa Euskadi, Arrasate / Mondragón, Basque Country, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia Oliveros I, Meabe Iturbe N, Marin Ojea JI, Lancho Poblador C, Fuentes-Claramonte P, Quemada Ubis JI. [Gross Motor Function after Rehabilitation with the Atlas 2030 Pediatric Exoskeleton in Children With Cerebral Palsy]. Rev Neurol. 2025 Aug 29;80(7):46141. doi: 10.31083/RN46141. Spanish. PMID 40916964